CLINICAL TRIAL: NCT07068906
Title: A Clinical Study to Investigate the Safety, Efficacy, and Cellular Metabolism of CT1194C CAR-T Cell Therapy, in Patients With Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: A Clinical Study Exploring CT1194C in Patients With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025069
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: B-Cell Non-Hodgkin Lymphoma
Keywords: CT1194C
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells chimeric antigen receptor T cells (Experimental)
  Interventions: Drug: CAR-T cells chimenric antigen receptor T cells

INTERVENTIONS:
Drug: CAR-T cells chimenric antigen receptor T cells — CT1194C cells infusion

SUMMARY:
A Clinical Study to Investigate the Safety, Efficacy, and Cellular Metabolism of CT1194C CAR-T Cell therapy, in Patients with Relapsed/Refractory B-Cell NonHodgkin Lymphoma.

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose exploratory clinical study to evaluate the safety, efficacy, cellular pharmacokinetics, and pharmacodynamics of CT1194C cells in patients with B-NHL. It is planned to enroll 3-27 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily sign the informed consent form (ICF) and must be willing and be able to adhere to the study visit schedule and other protocol requirements
2. 18-75 years old;
3. Histologically or cytologically confirmed B-NHL;
4. Previously received at least 2 lines of systemic therapy;
5. Intolerance to last treatment, or have progressed on or after the last treatment and currently require therapy;
6. There are measurable target lesions;
7. Expected survival > 12 weeks;
8. Eastern Cooperative Oncology Group (ECOG) score 0-1;
9. Female participants of childbearing potential must have a negative pregnancy test at screening and prior to receiving preconditioning therapy。Both male and Female are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment and are absolutely prohibited from donating sperm donation or eggs for 1 year after receiving study treatment infusion during the study;

Exclusion Criteria:

1. Pregnant or lactating women;
2. Has HIV, syphilis infection, active hepatitis B virus infection (HBsAg positive and HBV-DNA above the detection limit), or active hepatitis C virus infection (HCV antibody and HCV-DNA positive);
3. Has any current uncontrolled active infection, including but not limited to participants with active tuberculosis (investigator 's judgment);
4. Participants' toxicities caused by previous treatment did not recover to Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade 1, except alopecia and other events that are judged tolerable by the investigator;
5. Has received treatment for the disease within 14 days before informed consent, including but not limited to cytotoxic therapy, monoclonal antibodies or ADCs, targeted therapy, radiotherapy, epigenetic therapy, or investigational agents, or invasive investigational medical devices within 14 days before informed consent. If the radiation field covers ≤ 5% of the bone marrow reserve, the participant is eligible regardless of the end date of radiotherapy;
6. Systemic glucocorticoids equivalent to > 15 mg/day prednisone within 7 days prior to informed consent, with the exception of topical glucocorticoids;
7. Vaccination with live attenuated vaccines, inactivate vaccines or RNA vaccines within 4 weeks prior to informed consent;
8. Participants who are allergic or intolerant to preconditioning drugs, tocilizumab, or have other previous history of severe allergy such as anaphylactic shock;
9. Patients with any heart disease in the 6 months prior to screening;
10. Oxygen saturation < 92%,;
11. Presence of a second primary malignancy requiring treatment or not in complete remission within the past 2 years;
12. Major surgery within 2 weeks before informed consent or planned during the study period or within 4 weeks after giving study treatment (excluding local anesthesia such as cataract);
13. Participants are unable or unwilling to comply with the requirements of the study protocol or are otherwise unsuitable for participating in this clinical study in the investigator 's assessment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) after CT1194C infusion | 12 months after CT1194C infusion
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria
MTD and/or dose range | Up to 28 days after CAR-T cells infusion
  Evaluate Dose limited toxicity and recommended dosage range after CT1194C infusion

SECONDARY OUTCOMES:
Overall response rate （ORR） | Evaluate at 4, 8, 12 weeks and 6,9,12month after CAR-T infusion
  The proportion of patients with complete remission（CR）/partial response (PR) after CT1194C infusion.
Complete response rate (CRR) | 12 months after CT1194C infusion
  The proportion of patients with complete response(CR) after CT1194C infusion
Duration of remission(DOR) | 12 months after CT1194C infusion
  Participants achieving CR/PR will be included in the analysis set for DOR. DOR is defined as the time from the date of confirmed response until the date of disease relapse or death from any cause, whichever occurs first.
Time to response (TTR) | 12 months after CT1194C infusion
  The time from cell infusion to the first assessment of CR or PR
Time to complete response (TTCR) | 12 months after CT1194C infusion
  The time from cell infusion to the first assessment of CR
Progression-free survival (PFS) | 12 months after CT1194C infusion
  The time from the infusion of CT1194C cells to the first assessment of disease progression or death.
Overall survival (OS) | 12 months after CT1194C infusion]
  defined as the time from the date of receiving the infusion to the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- China Institute of Hematology and Blood Diseases Hospital, Tianjin, China